CLINICAL TRIAL: NCT06706999
Title: Pilot Study of Feasibility and Acceptability of PREVAIL (PREserving Valued Activities In Life)
Brief Title: Feasibility and Acceptability of PREVAIL (PREserving Valued Activities In Life)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-1195; 1K23AR079037 (NIH)
Record Dates: First submitted 2024-11-22; First posted 2024-11-27 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis (RA); Arthritis, Rheumatoid (RA)
Keywords: Physical Therapy; Rehabilitation
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants will all receive a recommendation from their rheumatology provider based on their DAPS score. Recommendations will consist of an exercise resource and potentially a referral for a brief PT consultation call.
  Interventions: Other: PREVAIL model of care

INTERVENTIONS:
Other: PREVAIL model of care — Components 1, 2, and 3 are essential components that all participants will receive. Components 4 and 5 are based on the results of either the DAPS tool or the PT consultation call.
  1. Screening tool (DAPS) completed at baseline to determine current level of limitation with valued life activities.
  2. Recommendation to rheumatology clinician based on screening results to provide exercise resource and/or recommend a PT consult call during routine visit.
  3. Exercise resource (PREVAIL website) provided to all participants by their rheumatology clinician at their routine visit.
  4. Brief consultation call with a study physical therapist to determine level of priority for PT referral. Only applicable for those with/at risk for limitation with valued life activities.
  5. Referral to PT. Only applicable if determined by study physical therapist to meet priority requirements.

SUMMARY:
The goal of this clinical trial is to learn if the PREVAIL model of care is a feasible way to integrate rehabilitation into routine rheumatology care for adults with rheumatoid arthritis (RA). The model of care consists of three essential components: a screening tool (Daily Activity and Participation Screen (DAPS)), a recommendation to the rheumatology clinician regarding rehabilitation referral and exercise, and an online exercise resource tailored for adults with RA.

Participants will complete baseline assessments before their scheduled routine visit with a rheumatology clinician, attend their visit, receive their exercise and/or rehabilitation recommendation, and complete follow-up assessments roughly three months after their visit. Based on a participant's DAPS score, they may be recommended to complete a brief consultation call with a study physical therapist, who may or may not refer them to physical therapy (PT). Participants may also be asked to elaborate on their experience with the PREVAIL model of care in an interview.

DETAILED DESCRIPTION:
Physical therapy and exercise interventions reduce impairment by improving pain, weakness, and fatigue. Despite continued high prevalence of functional limitations, often related to pain, weakness, and/or fatigue, PT and exercise are underutilized for adults with RA in the US. These low utilization rates do not align with the high impairment rate (up to 92%). Rheumatologists are without clear guidance regarding when to refer for PT, which may contribute to low utilization.

Physical activity and exercise are unequivocally beneficial for adults with RA, yet recommendations from providers are often limited, generic, or vague. Adults with RA have lower physical activity levels than the general population, including those with low symptom activity. Patients want information from a trusted expert who understands RA. Further, receiving a provider recommendation for exercise is strongly associated with engagement. Systematically integrating exercise recommendations, tailored to RA, in routine RA care is needed to increase exercise and delay limitations in discretionary activities.

The PREVAIL model of care was developed to preserve valued activities in life and facilitate the integration of PT for adults with RA who need it. The preliminary version of the PREVAIL model of care was developed based on current literature, which consistently identified a need for non-pharmacological treatment strategies for RA, and had three primary components: (1) Daily Activity and Participation Screening. Participants completed the S-VLA and were categorized into current level of limitation with valued life activities. This component was critical because there are currently no systematic methods to guide intervention in RA care in the US. (2) Recommendation for Referral to PT. The rheumatology clinician received a recommendation to refer to PT for patients with or at risk for limitation. (3). Exercise Guidance. All participants received evidence-based, RA-specific exercise guidance via web-based videos and links to self-directed and community resources that were developed and curated by previous research. This component was critical because exercise preserves function in adults with RA, and these patients want exercise guidance from trusted sources that acknowledge their RA.

This study builds on preparatory survey and interview studies to help refine the PREVAIL model of care before testing in this pilot clinical trial. The investigators have added an interim PT consultation call with a study physical therapist as the initial referral from the rheumatology clinician, and refined the timeline with which assessments are administered.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Clinician diagnosis of RA as defined by International Classification of Diseases 10 (ICD-10) code
* Receiving routine care from a UNC rheumatology clinician
* Have an upcoming scheduled visit with a UNC rheumatology clinician for a routine follow up

Exclusion Criteria:

* No documented diagnosis of RA
* Under the age of 18
* Significant cognitive impairment
* Condition that restricts ability to complete surveys and patient reported outcomes
* Severe hearing or visual impairment
* Serious/terminal illness as indicated by referral to hospice or palliative care
* Unable to speak or read English
* Current participation in any other study related to RA
* Current or recent (within the last six months) participation in PT
* Recent (within the last 6 months) major surgery requiring overnight hospital admission and/or resulting in functional loss, requiring rehabilitation
* Upcoming (within the next 6 months) major surgery requiring overnight hospital admission and/or resulting in functional loss, requiring rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-11-16 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who receive PREVAIL model of care essential components | Baseline assessments (including the DAPS tool) provided 1 week before routine visit, routine visit with rheumatology clinician, and 3-month follow-up assessments
  Data will be collected from participants and rheumatology clinicians on whether or not essential components were administered. This is necessary for assessing the feasibility of the PREVAIL model of care.
Percentage of participants who access the exercise resource at least once during study duration | Collected during 3-month follow-up assessments
  Exercise resource utilization will be measured through patient report and google analytics to determine feasibility of the PREVAIL model of care from the patient perspective.
Average score on the Feasibility of Intervention Measure (FIM) | Collected during 3-month follow-up assessments
  The FIM is a method for determining if a treatment or intervention can be carried out in a particular setting. It is a valid and reliable 4-item outcome measure scored on a 5-point Likert scale (completely disagree = 1, completely agree = 5). Higher scores indicate higher feasibility. This is essential for assessing the PREVAIL model of care from the patient perspective.
Average score on the Acceptability of Intervention Measure (AIM) | Collected during 3-month follow-up assessments
  The AIM is a valid and reliable 4-item outcome measure to test whether the intervention is agreeable and appealing to individuals. It is also scored on a 5-point Likert scale, with higher answers indicating higher acceptability. AIM scores will be used to assess the PREVAIL model of care from the patient perspective.

SECONDARY OUTCOMES:
Percentage of recruitment pool who enroll in the study | EMR Review and Pre-Screening (2 months prior to appointment) to enrollment (2 months to 1 week before routine visit)
  The percentage of recruitment pool who pass electronic medical record (EMR) chart review and study pre-screening, then proceed to enroll in the study will be collected. This is essential for assessing the feasibility of conducting a larger scale trial of the PREVAIL model of care.
Percentage of participants that complete follow-up assessments | Assessments provided 3 months after baseline assessment visit
  The study team will track completion of each assessment through REDCap. This is necessary for determining the feasibility of a larger scale trial of the PREVAIL model of care.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Thoma, DPT, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

DOCUMENTS (1):
  • Informed Consent Form (2025-05-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT06706999/ICF_000.pdf